CLINICAL TRIAL: NCT05867797
Title: Risk Factors and Outcomes of Acute Kidney Injury in Patients With Diabetic Ketoacidosis at Sohag University Hospital.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Zahraa Abdelaal Ahmed, Internal medicine specialist, Sohag University
Other Study IDs: Soh-Med-23-05-03MD
Record Dates: First submitted 2023-05-10; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Diabetic Ketoacidosis; Acute Kidney Injury
Keywords: DKA AKI
MeSH Terms: conditions — Diabetic Ketoacidosis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood sample, urine sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Diabetic ketoacidosis (DKA), a severe complication of diabetes mellitus (DM), is the leading cause of hospitalization, morbidity and mortality in patients with DM (1).

DKA is associated with hyperglycemic crises and featured by metabolic acidosis, the production of ketoacids, volume depletion, and electrolyte imbalance. Due to glucose-induced osmotic polyuria and even emesis, volume depletion is a major cause of acute kidney injury (AKI) in DKA patients (2).

ELIGIBILITY:
Inclusion Criteria:

* patients will be included in this study aged >18 years old after diagnosis of AKI on top of Diabetic ketoacidosis at Sohag university hospital for all patients admitted during the period from May 2023 to May 2024

Exclusion Criteria:

* Chronic kidney disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic ketoacidosis at Sohag university hospital for all patients admitted during the period from May 2023 to May 2024
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-20 (Estimated); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
prognosis risk factors and outcomes of AKI in patients with DKA | 1 YEAR
  complete resolution or progress to CKD or mortality and discover risk factors for AKI as uncontrolled diabetes infection or high uric acid uncontrolled hyperlipidemia